CLINICAL TRIAL: NCT04528979
Title: The Outcome of Endodontic Treatment and Retreatment With a Bioceramic Sealer: A Prospective Randomized Controlled Clinical Study
Brief Title: Outcome of Endodontic Treatment and Retreatment With a Bioceramic Sealer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juan Gonzalo Olivieri (Other)
Responsible Party: Sponsor-Investigator, Juan Gonzalo Olivieri, Principal investigator, Universitat Internacional de Catalunya
Organization: Universitat Internacional de Catalunya (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UICENDECL201703
Record Dates: First submitted 2020-05-21; First posted 2020-08-27 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Endodontic Disease; Endodontically Treated Teeth
Keywords: Primary root canal treatment; Secondary root canal treatment; Outcome; Root canal sealer
MeSH Terms: conditions — Dental Pulp Diseases; Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary root canal treatment (Experimental): Primary root canal treatment sealed with guttapercha and AH Plus® or BioRoot RCS® root canal sealers
  Interventions: Other: BioRoot RCS® root canal sealer; Other: AH Plus® root canal sealer
- Secondary root canal treatment (Experimental): Secondary root canal treatment sealed with guttapercha and AH Plus® or BioRoot RCS® root canal sealers
  Interventions: Other: BioRoot RCS® root canal sealer; Other: AH Plus® root canal sealer

INTERVENTIONS:
Other: BioRoot RCS® root canal sealer — Root canal obturation with guttapercha and BioRoot RCS® root canal sealer
Other: AH Plus® root canal sealer — Root canal obturation with guttapercha and AH Plus® root canal sealer

SUMMARY:
This study is a prospective randomized controlled study of patients who come to the University. The aim is to evaluate the success rate of treatment and retreatment of canals using BioRoot ™ RCS cement compared with AH Plus up to 6 years of follow-up. The null hypothesis is that there will be no statistically significant differences in rates of successful treatment of root canals filled with BioRoot ™ RCS compared to gutta-percha and AH Plus sealer.

ELIGIBILITY:
Inclusion Criteria:

* Patients that demonstrate understanding of the study and willingness to participate as evidenced by signing the voluntary informed consent and received a signed and dated copy of the informed consent form.
* Understands and is willing to comply with all study procedures and restrictions.
* Not presence of clinically significant and relevant abnormalities of clinical history or oral examination.
* Diagnosis of irreversible pulpitis or apical symptomatic / asymptomatic periodontitis.
* Retreatment cases due to an endodontic failure.
* Single or bi-radicular teeth.

Exclusion Criteria:

* General: Patients with systemic diseases, diabetes, immunocompromised and pregnant women, or any clinically significant or relevant oral abnormalities.
* Specific: root resorption, root fractures, impossibility of restoration and cases were primary or secondary root canal treatment is not the treatment of choice.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Clinical post-operative pain | Immediately post-treatment.
  VAS score of patient' level of pain, from no pain to extreme pain
Clinical post-operative pain | 4 hours post-treatment
  VAS score of patient' level of pain, from no pain to extreme pain
Clinical post-operative pain | 24 hours post treatment
  VAS score of patient' level of pain, from no pain to extreme pain
Clinical post-operative pain | 48 hours post treatment
  VAS score of patient' level of pain, from no pain to extreme pain
Clinical signs or symptoms of periapical disease | 1 year
  Absence/presence of clinical signs or symptoms of periapical disease
Clinical signs or symptoms of periapical disease | 2 years
  Absence/presence of clinical signs or symptoms of periapical disease
Clinical signs or symptoms of periapical disease | 4 years
  Absence/presence of clinical signs or symptoms of periapical disease
Clinical signs or symptoms of periapical disease | 6 years
  Absence/presence of clinical signs or symptoms of periapical disease
Radiographic periapical healing | 1 year
  Absence/presence of radiographic apical periodontitis + PAI changes when compared with post-treatment radiograph
Radiographic periapical healing | 2 years
  Absence/presence of radiographic apical periodontitis + PAI changes when compared with post-treatment radiograph
Radiographic periapical healing | 4 years
  Absence/presence of radiographic apical periodontitis + PAI changes when compared with post-treatment radiograph
Radiographic periapical healing | 6 years
  Absence/presence of radiographic apical periodontitis + PAI changes when compared with post-treatment radiograph

SECONDARY OUTCOMES:
Correlation of prognostic factors and clinical signs or symptoms of periapical disease | 1 year
  Correlation of Pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist with having clinical signs or symptoms of periapical disease
Correlation of prognostic factors and clinical signs or symptoms of periapical disease | 2 years
  Correlation of Pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist with having clinical signs or symptoms of periapical disease
Correlation of prognostic factors and clinical signs or symptoms of periapical disease | 4 years
  Correlation of Pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist with having clinical signs or symptoms of periapical disease
Correlation of prognostic factors and clinical signs or symptoms of periapical disease | 6 years
  Correlation of Pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist with having clinical signs or symptoms of periapical disease
Correlation of prognostic factors and radiographic periapical healing | 1 year
  Pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist, in relation to radiographic periapical Correlation of Pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist with radiographic periapical healing
Correlation of prognostic factors and radiographic periapical healing | 2 years
  Correlation of Pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist with radiographic periapical healing
Correlation of prognostic factors and radiographic periapical healing | 4 years
  Correlation of Pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist with radiographic periapical healing
Correlation of prognostic factors and radiographic periapical healing | 6 years
  Correlation of Pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist with radiographic periapical healing

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No